CLINICAL TRIAL: NCT00748618
Title: Vitamin D Replacement After Kidney Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0382-08-FB
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-08

CONDITIONS: Kidney Transplantation; Vitamin D Deficiency
Keywords: Kidney transplantation (KTX); Vitamin D deficiency; Cardiovascular Disease (CVD); Vascular risk; Parathyroid hormone (PTH); Carotid intima media thickness (CIMT); Insulin resistance (IR)
MeSH Terms: conditions — Vitamin D Deficiency; Cardiovascular Diseases; Insulin Resistance | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard vitamin treatment (Other): 10,000 I.U. of vitamin D3 weekly
  Interventions: Dietary Supplement: Standard vitamin D3 treatment
- 50,000 I.U. of vitamin D3 (Active Comparator): 50,000 I.U. of vitamin D3 weekly
  Interventions: Dietary Supplement: High dose vitamin D3 treatment

INTERVENTIONS:
Dietary Supplement: Standard vitamin D3 treatment — 10,000 I.U./wk of vitamin D3 orally for 6 months
  Arms: Standard vitamin treatment
Dietary Supplement: High dose vitamin D3 treatment — 50,000 I.U./wk of vitamin D3 orally for 6 months
  Other Names: D3, vitamin D
  Arms: 50,000 I.U. of vitamin D3

SUMMARY:
Vitamin D deficiency accelerates vascular risk progression after kidney transplant.

DETAILED DESCRIPTION:
This trial will assess the following aims:

1. Time to plateau vitamin D concentrations after initiating vitamin D supplements
2. Safety of vitamin D replacement based on serum and urine calcium
3. Effect of vitamin D on PTH concentration in individuals with elevated parathyroid hormone
4. Effect of vitamin D on markers of insulin resistance and inflammation

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant more than 6 months ago
* 19 years or older
* 25-hydroxy vitamin D ≤35 ng/ml

Exclusion Criteria:

* Estimated Glomerular filtration rate (GFR) <30 ml/min/1.73m²
* Previous small bowel or lung transplant
* Pancreas transplant less than 6 months ago
* Cancer or any condition that would change their weight dramatically in the near future such as malabsorption
* Willing to return for testing every two months
* Women who are pregnant or < 6 weeks postpartum
* Calcium > 10.5 mg/dl
* Phosphate > 4.8 mg/dl
* Drinking more than 2 alcohol drinks a day or 14 drinks per week
* History of parathyroid surgery
* Known granulomatous disease
* Taking any seizure medication that affects vitamin D
* Taking Zemplar ® and/or Rocaltrol ®
* History of kidney stones in the past 20 years
* Not on a stable dose of bisphosphonate for the past three months
* Planning on a pancreas transplant within the next year
* In any other research study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2012-04-01 (Actual); Study Completion 2023-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Larsen, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 165 subjects were screened, and 93 subjects were eligible and were randomized to treatments. Three patients voluntarily withdrew consent immediately following randomization. A total of 90 subjects received treatments.
Groups:
- Standard Vitamin Treatment: Standard vitamin treatment
  vitamin D3: Participants receive 10,000 I.U./wk of vitamin D3 orally for 6 months
- 50,000 I.U. of Vitamin D3: 50,000 I.U. of vitamin D3
  vitamin D3: Participants receive 50,000 I.U./wk of vitamin D3 orally for 6 months
Period: Overall Study
Arm/Group | Standard Vitamin Treatment | 50,000 I.U. of Vitamin D3
Started | 46 | 44
Completed | 45 | 44
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Vitamin Treatment: Standard vitamin treatment
  vitamin D3: 10,000 I.U./wk of vitamin D3 orally for 6 months
- 50,000 I.U. of Vitamin D3: 50,000 I.U. of vitamin D3
  vitamin D3: 50,000 I.U./wk of vitamin D3 orally for 6 months
- Total: Total of all reporting groups
Arm/Group | Standard Vitamin Treatment | 50,000 I.U. of Vitamin D3 | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (10.5) | 52.1 (12.1) | 53.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 21 | 48
  Male | 19 | 23 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 43 | 40 | 83
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 40 | 37 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Vitamin D Concentration [Mean (Standard Deviation); unit: ng/ml] | 27.2 (5.3) | 26.3 (6.9) | 26.7 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Compare Efficacy and Safety of Two Vitamin D Supplements of These Doses in Normalizing Vitamin D Concentrations.
Description: The 6 month change (6 month - Baseline) was compared between the two treatment arms of vitamin D supplements for normalizing vitamin D concentrations. Higher change values indicate improvement in vitamin D levels.
Time Frame: Baseline and 6 months
Population: Patients who had baseline and 6 month 25-hydroxy Vitamin D levels measured
Measure: Median (Full Range); unit: ng/ml
Arm/Group | Standard Vitamin Treatment | 50,000 I.U. of Vitamin D3
Number analyzed (Participants) | 45 | 43
ng/ml | 8 [-10 to 32] | 29 [-9 to 61]

2. Secondary Outcome: The Ability of Vitamin D to Reduce Parathyroid Hormone Concentration.
Description: The 6 month change (6 month - Baseline) in parathyroid hormone concentration was compared between the two treatment arms.
Time Frame: baseline and 6 months
Population: Available data from patients who had baseline and 6 month parathyroid hormone concentration levels obtained.
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Standard Vitamin Treatment | 50,000 I.U. of Vitamin D3
Number analyzed (Participants) | 45 | 43
pg/ml | 1.0 [-120.6 to 81.0] | -9.0 [-94.0 to 200.0]

3. Secondary Outcome: The Ability of Vitamin D to Alter Spot Urine Protein-Creatinine Ratio.
Description: The 6 month change (6 month - Baseline) in spot urine protein-creatinine ratio was compared between the two treatment arms.
Time Frame: 6 months
Population: Available data from patients who had baseline and 6 month spot urine protein-creatinine ratio levels obtained.
Measure: Median (Full Range); unit: mg/mmol
Arm/Group | Standard Vitamin Treatment | 50,000 I.U. of Vitamin D3
Number analyzed (Participants) | 44 | 42
mg/mmol | -0.45 [-1215.4 to 1906.7] | -1.95 [-1652.7 to 798.8]

4. Secondary Outcome: The Effect of Vitamin D Supplementation on 6 Month High-sensitivity C-reactive Protein (HsCRP) Levels.
Description: The 6 month change in High-sensitivity C-reactive protein (HsCRP) levels was compared between the two treatment arms.
Time Frame: Baseline and 6 months
Population: Available data from patients who had baseline and 6 month HsCRP levels obtained
Measure: Median (Full Range); unit: mg/dl
Arm/Group | Standard Vitamin Treatment | 50,000 I.U. of Vitamin D3
Number analyzed (Participants) | 45 | 42
mg/dl | 0.3 [-13.5 to 18.4] | 0.15 [-42.2 to 51.3]

5. Secondary Outcome: The Effect of Vitamin D Supplementation on Insulin Resistance at 6 Months
Description: The 6 month change (6 month - Baseline) in insulin resistance was assessed with HOMA-IR (Homeostatic Model Assessment-Insulin Resistance), which is calculated by fasting glucose (mg/dL) X fasting insulin (mU/L) /405.
Time Frame: Baseline and 6 months
Population: Available data from patients who had baseline and 6 month HOMA-IR levels obtained.
Measure: Median (Full Range); unit: (microU/L) x (nmol/L)
Arm/Group | Standard Vitamin Treatment | 50,000 I.U. of Vitamin D3
Number analyzed (Participants) | 30 | 26
(microU/L) x (nmol/L) | -0.6 [-7.2 to 4.3] | 0.1 [-7.0 to 8.0]

ADVERSE EVENTS:
Arm/Group | Standard Vitamin Treatment | 50,000 I.U. of Vitamin D3
Serious Adverse Events (participants affected / at risk) | 0/46 | 1/44
Other Adverse Events (participants affected / at risk) | 1/46 | 2/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Vitamin Treatment (N=46) | 50,000 I.U. of Vitamin D3 (N=44)
Viral gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reoccurring UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
Enteric Conversion (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Vitamin Treatment (N=46) | 50,000 I.U. of Vitamin D3 (N=44)
Elevated calcium (Endocrine disorders) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes